CLINICAL TRIAL: NCT00261898
Title: Chronic Sleep Deprivation as a Risk Factor for Metabolic Syndrome and Obesity
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study has been terminated. (Interim analysis of preliminary results indicated the need for protocol re-design).
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060036; 06-DK-0036
Record Dates: First submitted 2005-12-04; First posted 2005-12-05 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Obesity; Chronic Sleep Deprivation
Keywords: Sleep Deprivation; Obesity; Metabolic Syndrome; Hormones; Public Health; Overweight; Sleep
MeSH Terms: conditions — Obesity; Sleep Deprivation; Metabolic Syndrome; Overweight

INTERVENTIONS:
Procedure: Increase sleep

SUMMARY:
OBJECTIVE: Obesity and chronic sleep deprivation have both become increasingly pervasive medical problems in recent years. The prevalence of adult obesity has doubled over the past 30 years and continues to increase. In addition, industrial societies attach an economic value to maximizing the waking period to the longest tolerable limit by sleeping as little as possible. Average sleep time has decreased over the last century by 2 hours. Chronically sleeping less has been associated with increased weight, endocrine and metabolic health risks including glucose intolerance, cardiovascular disease, and mortality. The possibility that the current epidemic of obesity and metabolic health risks may be partially related to insufficient sleep is now being recognized. The objective of this proof-of-concept controlled trial is to investigate the impact of increasing sleep time in chronically sleep-deprived, obese subjects.

STUDY POPULATION: 18-50 year old, obese (BMI 30-50) men and premenopausal women, chronically sleep deprived, recruited from the Baltimore-Washington metropolitan area. Chronic sleep deprivation will be verified by the use of sleep logs and the use of actigraphy before entry into the study. Secondary causes of sleep deprivation such as insomnia, psychological (depression), and medical conditions associated with poor sleep quality (including obstructive sleep apnea) will be exclusionary criteria.

DESIGN: This is a randomized, 12-month duration, comparison-controlled clinical trial of an extension of sleep up to approximately 7 hours and 30 minutes (Intervention Group) or continuation of habitual short sleep schedule (Comparison Group). The proposed treatment is an educational and behavioral intervention aimed at increasing sleep in a non-pharmacological fashion. The main analysis of the study will be to determine if additional sleep will result in a significant difference in body weight at the end of 12 months between the Intervention Group and the Comparison Group. In addition, we would like to establish whether 12 months of additional sleep will result in: a) a decreased prevalence of metabolic syndrome; and b) changes in the endocrine profile (i.e. inducing changes in leptin [increase] and ghrelin [decrease] opposite to the changes associated with chronic sleep deprivation). At the end of the 12-month intervention study (Phase 1, Efficacy Randomized Phase Study), all participants will be given information about the potential benefit of more sleep and encouraged to increase sleep time. Health teaching about proper nutrition and adequate exercise will also be provided at that time to the Intervention and Comparison Groups. All participants will be evaluated 6 months later to assess the effects of this intervention in a real-life situation, and offered participation in a three-year extension with semi-annual visits (Phase 2, Effectiveness 3 Year Follow-Up Phase Study), for which matched external comparison subjects will also be recruited ad hoc.

OUTCOME PARAMETERS: body weight, average number of hours of sleep/night, fasting glucose and insulin, oral glucose tolerance test, leptin, ghrelin, adiponectin, other relevant endocrine and anthropometric measures, body composition, various metabolic parameters, food intake, energy expenditure, and quality of life measures.

DETAILED DESCRIPTION:
OBJECTIVE: Obesity and chronic sleep deprivation have both become increasingly pervasive medical problems in recent years. The prevalence of adult obesity has doubled over the past 30 years and continues to increase. In addition, industrial societies attach an economic value to maximizing the waking period to the longest tolerable limit by sleeping as little as possible. Average sleep time has decreased over the last century by 2 hours. Chronically sleeping less has been associated with increased weight, endocrine and metabolic health risks including glucose intolerance, cardiovascular disease, and mortality. The possibility that the current epidemic of obesity and metabolic health risks may be partially related to insufficient sleep is now being recognized. The objective of this proof-of-concept controlled trial is to investigate the impact of increasing sleep time in chronically sleep-deprived, obese subjects.

STUDY POPULATION: 18-50 year old, obese (BMI 29-55) men and premenopausal women, chronically sleep deprived, recruited from the Baltimore-Washington metropolitan area. Chronic sleep deprivation will be verified by the use of sleep logs and the use of actigraphy before entry into the study. Secondary causes of sleep deprivation such as insomnia, psychological (depression), and medical conditions associated with poor sleep quality (including obstructive sleep apnea) will be exclusionary criteria.

DESIGN: This is a randomized, 12-month duration, comparison-controlled clinical trial of an extension of sleep up to approximately 7 hours and 30 minutes (Intervention Group) or continuation of habitual short sleep schedule (Comparison Group). The proposed treatment is an educational and behavioral intervention aimed at increasing sleep in a non-pharmacological fashion. The main analysis of the study will be to determine if additional sleep will result in a significant difference in body weight at the end of 12 months between the Intervention Group and the Comparison Group. In addition, we would like to establish whether 12 months of additional sleep will result in: a) a decreased prevalence of metabolic syndrome; and b) changes in the endocrine profile (i.e. inducing changes in leptin [increase] and ghrelin [decrease] opposite to the changes associated with chronic sleep deprivation). At the end of the 12-month intervention study (Phase 1, Efficacy [Randomized Phase] Study), all participants will be given information about the potential benefit of more sleep and encouraged to increase sleep time. Health teaching about proper nutrition and adequate exercise will also be provided at that time to the Intervention and Comparison Groups. All participants will be evaluated 6 months later to assess the effects of this intervention in a real-life situation, and offered participation in a three-year extension with semi-annual visits (Phase 2, Effectiveness [3 Year Follow-Up Phase] Study), for which matched external comparison subjects will also be recruited ad hoc.

OUTCOME PARAMETERS: body weight, average number of hours of sleep/night, fasting glucose and insulin, oral glucose tolerance test, leptin, ghrelin, adiponectin, other relevant endocrine and anthropometric measures, body composition, various metabolic parameters, food intake, energy expenditure, and quality of life measures.

The study was terminated early for reasons of apparent futility of continuing accrual of participants according to the original study plan. The decision was based on independent analysis of data acquired during the initial feasibility phase and from interim analysis of early results that failed to document objectively the achievement of substantive and meaningful differences between experimental and control groups with respect to amounts of sleep extension, changes in metabolic parameters, or changes in weight. Feasibilities of achieving objective and substantive differences in these parameters were integral to the methodology of the original study plan and required to meet the statistical power calculations for the controlled trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

  18 to 50 year old obese men and premenopausal women

BMI between 29-55

Chronically (for more than 6 months) sleep-deprived, defined as sleeping on a regular basis less than or equal to approximately 6-1/2 hours/night by history and objective devices (wrist activity monitors and sleep logs).

INCLUSION CRITERIA: External comparison subjects for extension of Effectiveness Study must meet the criteria above.

EXCLUSION CRITERIA:

Diagnosed sleep disorders including:

* Chronic insomnia
* Untreated sleep disordered breathing (sleep apnea at a level of severity [using standardized criteria for measurement], or diagnosed UARS [upper airway resistance syndrome] that would impair the ability to increase sleep duration [Intervention Group] or maintain sleep duration [Comparison Group]. CPAP treatment that has been in place for 3 months or more and improves sleep is acceptable).
* Restless leg syndrome or periodic limb movement disorder
* Parasomnias (including REM sleep behavior disorders, confusional arousals, sleep terrors, sleepwalking, sleep violence)
* Primary bruxism is allowed as long as it does not interfere with the ability to sleep an additional 90 minutes a night
* Narcolepsy
* Central apnea.

Unstable weight (voluntary losses in BMI greater than 5% over the past 6 months); currently being enrolled in a weight loss program

Untreated or uncontrolled diabetes

Severe uncontrolled hypertension

Other chronic organ disease diagnosis including:

* COPD
* Chronic cardiac arrhythmia requiring treatments
* Gastro-esophageal disorders associated with sleep-related symptoms.

Medications

* chronic use of prescription or over-the-counter medications known to affect sleep (e.g., systemic steroids, NSAIDs)
* current anticonvulsant therapy

Chronic fatigue syndrome and fibromyalgia

Acromegaly, hypothyroidism (unless on a stable replacement dose of thyroid hormone), Cushing disease or other endocrine disorders known to affect sleep

Poorly controlled major depression (subjects who have been on a stable pharmacological antidepressant treatment for 3 months and are in remission without substantial weight gain are eligible).

Other current DSM-IV diagnoses, including:

* Eating disorders such as bulimia nervosa and binge eating disorder
* Anxiety disorders such as PTSD and panic attacks
* Mania
* Schizophrenia.

Medication and substance abuse such as excessive alcohol consumption or drug abuse or dependence that may pose a threat to compliance

Being a rotating worker, shift worker (working evenings or nights), or long distance commuter (more than approximately 90 minutes each way), traveling frequently outside of time zone; being in an occupation that may require special vigilance such as driving a truck, bus, or cab; operating heavy machinery; being a pilot or air traffic controller

Being likely to move to a different geographical area during the study

Having a sleep partner that would make compliance with study requirements difficult

Pregnancy and lactation

Menopause

Chronic excessive caffeine use (habitual intake of more than 500 mg/day)

Any condition that in the opinion of the principal investigator makes study participation and compliance problematic.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 239 (Actual)
Dates: Start 2005-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Cizza, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cizza G, Skarulis M, Mignot E. A link between short sleep and obesity: building the evidence for causation. Sleep. 2005 Oct;28(10):1217-20. doi: 10.1093/sleep/28.10.1217. No abstract available. PMID 16295203
- [Background] Cizza G, Romagni P, Lotsikas A, Lam G, Rosenthal NE, Chrousos GP. Plasma leptin in men and women with seasonal affective disorder and in healthy matched controls. Horm Metab Res. 2005 Jan;37(1):45-8. doi: 10.1055/s-2005-861033. PMID 15702439
- [Background] Bray GA. Medical consequences of obesity. J Clin Endocrinol Metab. 2004 Jun;89(6):2583-9. doi: 10.1210/jc.2004-0535. PMID 15181027
- [Background] Gangwisch JE, Malaspina D, Boden-Albala B, Heymsfield SB. Inadequate sleep as a risk factor for obesity: analyses of the NHANES I. Sleep. 2005 Oct;28(10):1289-96. doi: 10.1093/sleep/28.10.1289. PMID 16295214
- [Background] Hasler G, Buysse DJ, Klaghofer R, Gamma A, Ajdacic V, Eich D, Rossler W, Angst J. The association between short sleep duration and obesity in young adults: a 13-year prospective study. Sleep. 2004 Jun 15;27(4):661-6. doi: 10.1093/sleep/27.4.661. PMID 15283000
- [Background] Spiegel K, Tasali E, Penev P, Van Cauter E. Brief communication: Sleep curtailment in healthy young men is associated with decreased leptin levels, elevated ghrelin levels, and increased hunger and appetite. Ann Intern Med. 2004 Dec 7;141(11):846-50. doi: 10.7326/0003-4819-141-11-200412070-00008. PMID 15583226
- [Background] Wehr TA. Effect of seasonal changes in daylength on human neuroendocrine function. Horm Res. 1998;49(3-4):118-24. doi: 10.1159/000023157. PMID 9550111
- [Background] Cizza G, Piaggi P, Rother KI, Csako G; Sleep Extension Study Group. Hawthorne effect with transient behavioral and biochemical changes in a randomized controlled sleep extension trial of chronically short-sleeping obese adults: implications for the design and interpretation of clinical studies. PLoS One. 2014 Aug 20;9(8):e104176. doi: 10.1371/journal.pone.0104176. eCollection 2014. PMID 25141012
- [Background] Cizza G, Marincola P, Mattingly M, Williams L, Mitler M, Skarulis M, Csako G. Treatment of obesity with extension of sleep duration: a randomized, prospective, controlled trial. Clin Trials. 2010 Jun;7(3):274-85. doi: 10.1177/1740774510368298. Epub 2010 Apr 27. PMID 20423926
- [Derived] Lucassen EA, Piaggi P, Dsurney J, de Jonge L, Zhao XC, Mattingly MS, Ramer A, Gershengorn J, Csako G, Cizza G; Sleep Extension Study Group. Sleep extension improves neurocognitive functions in chronically sleep-deprived obese individuals. PLoS One. 2014 Jan 15;9(1):e84832. doi: 10.1371/journal.pone.0084832. eCollection 2014. PMID 24482677
- [Derived] Cizza G, Piaggi P, Lucassen EA, de Jonge L, Walter M, Mattingly MS, Kalish H, Csako G, Rother KI; Sleep Extension Study Group. Obstructive sleep apnea is a predictor of abnormal glucose metabolism in chronically sleep deprived obese adults. PLoS One. 2013 May 29;8(5):e65400. doi: 10.1371/journal.pone.0065400. Print 2013. PMID 23734252
- [Derived] Lucassen EA, Zhao X, Rother KI, Mattingly MS, Courville AB, de Jonge L, Csako G, Cizza G; Sleep Extension Study Group. Evening chronotype is associated with changes in eating behavior, more sleep apnea, and increased stress hormones in short sleeping obese individuals. PLoS One. 2013;8(3):e56519. doi: 10.1371/journal.pone.0056519. Epub 2013 Mar 6. PMID 23483886
- [Derived] de Jonge L, Zhao X, Mattingly MS, Zuber SM, Piaggi P, Csako G, Cizza G; NIDDK Sleep Extension Study Group. Poor sleep quality and sleep apnea are associated with higher resting energy expenditure in obese individuals with short sleep duration. J Clin Endocrinol Metab. 2012 Aug;97(8):2881-9. doi: 10.1210/jc.2011-2858. Epub 2012 Jun 11. PMID 22689694
- [Derived] Knutson KL, Galli G, Zhao X, Mattingly M, Cizza G; NIDDK Sleep Extension Study. No association between leptin levels and sleep duration or quality in obese adults. Obesity (Silver Spring). 2011 Dec;19(12):2433-5. doi: 10.1038/oby.2011.248. Epub 2011 Jul 28. PMID 21799479